CLINICAL TRIAL: NCT05028361
Title: Safety of Simultaneous Versus Sequential Administration of mRNA COVID-19 Vaccines and Quadrivalent Inactivated Influenza (IIV4) in Adults, Adolescents and Children: A Randomized Observer Blinded Study
Brief Title: Simultaneous mRNA COVID-19 and IIV4 Vaccination Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Johns Hopkins University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00109102
Record Dates: First submitted 2021-08-30; First posted 2021-08-31 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Quality of Life; Injection Site Reaction; Adverse Drug Event; Systemic Reaction
Keywords: COVID-19; Influenza; vaccine; mRNA COVID-19 vaccine; influenza vaccine; safety; quality of life; pain following vaccination; fever following vaccination
MeSH Terms: conditions — Injection Site Reaction; Drug-Related Side Effects and Adverse Reactions; COVID-19; Influenza, Human | interventions — 2019-nCoV Vaccine mRNA-1273; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simultaneous Vaccination Group (Other): Subjects will receive a dose of mRNA COVID-19 vaccine (either as a study procedure or standard of care) and IIV4 at Visit 1, saline placebo at Visit 2, and mRNA COVID-19 vaccine at Visit 3 (only for participants receiving their primary series of mRNA COVID-19 vaccine.)
  Interventions: Biological: mRNA COVID-19; Biological: IIV4; Other: Placebo (saline)
- Sequential Vaccination Group (Other): Subjects will receive a dose of mRNA COVID-19 vaccine (either as a study procedure or standard of care) and saline placebo at Visit 1, IIV4 at Visit 2, and mRNA COVID-19 vaccine at Visit 3 (only for participants receiving their primary series of mRNA COVID-19 vaccine.)
  Interventions: Biological: mRNA COVID-19; Biological: IIV4; Other: Placebo (saline)

INTERVENTIONS:
Biological: mRNA COVID-19 — ACIP-CDC recommended vaccine
Biological: IIV4 — ACIP recommended vaccine
Other: Placebo (saline) — Saline Control

SUMMARY:
This study is a prospective, randomized clinical trial. During this study, participants will be randomly assigned to receive quadrivalent inactivated influenza vaccine (IIV4) and mRNA COVID-19 vaccine either simultaneously or sequentially, 7-14 days apart. Persons in the simultaneous group will receive mRNA COVID-19 and IIV4 at Visit 1 (Day 1) and a saline placebo injection at Visit 2. Persons in the sequential group will receive mRNA COVID-19 vaccine and a saline placebo at Visit 1 (Day 1) and IIV4 injection at Visit 2. For participants receiving their primary dose series, a second dose of mRNA COVID-19 vaccine will be administered either 3 to 8 weeks or 4 to 8 weeks following the first dose, depending upon the mRNA COVID-19 vaccine provided. For those receiving a booster dose of mRNA COVID-19 only a single mRNA COVID-19 will be received in this study. Solicited symptoms of reactogenicity and adverse events will be assessed on vaccination day and daily during the 7 days following each Vaccination Visit using either electronic or paper symptoms diaries, depending on study participant preference. Quality of life data will be collected using electronic or paper diaries on day of Vaccination Visit 1 and daily during the 7 days following the visit. Serious adverse events and adverse events of special interest will be collected throughout the duration of the study. Participants are followed through Day 121. Serum samples from participants will be collected for determination of SARS-CoV-2 seropositivity at baseline. Serum samples will be taken throughout the study to determine IIV4 and COVID-19 vaccine immunogenicity and for potential future studies.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged ≥5 years if receiving primary two-dose mRNA COVID-19 vaccine series or persons aged ≥12 years if receiving a booster mRNA COVID-19 vaccine dose according to FDA authorization or approval and ACIP recommendation. Note: receipt of an mRNA COVID-19 vaccine within 8 hours of enrollment is permitted

  *Individuals age 5-11 receiving a booster may be enrolled in the event a booster for individuals age 5-11 is authorized or approved and recommended by the ACIP.
* English or Spanish literate
* Intention of receiving influenza vaccine and COVID-19 vaccine based on ACIP-CDC guidelines
* Willing to provide written informed consent
* Intention of being available for entire study period and complete all relevant study procedures, including follow-up phone calls and clinic visits

Exclusion Criteria:

* Currently pregnant, planning to become pregnant within the first three months of the study per participant self-report or likely to be pregnant per screening criteria as defined in Section 5.1 at Visit 1
* Prior receipt of IIV4 during the respective influenza season in which they are being enrolled
* <9 years of age and recommended to receive two doses of IIV4 during the respective influenza season in which they are being enrolled
* Prior receipt of non-mRNA COVID-19 vaccine
* Documented COVID-19 infection within 6 weeks prior to enrollment confirmed by either medical history or lab testing
* History of severe allergic reaction after a previous dose of any influenza vaccine; or to an influenza vaccine component, including egg protein
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of an mRNA vaccine
* Receipt of any licensed inactivated vaccine within 2 weeks prior to enrollment in this study, receipt of any licensed live vaccine within 4 weeks prior to enrollment in this study, or receipt of Shingrix (Zoster Vaccine Recombinant, Adjuvanted) or HEPLISAV-B (Hepatitis B Vaccine (Recombinant), Adjuvanted) vaccine within 6 weeks prior to enrollment in this study or planning receipt of any vaccines following enrollment until 6 weeks after receipt of the second dose of mRNA COVID-19 vaccine
* Has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematologic malignancy* *Participants with a history of malignancy may be included if, after previous treatment by surgical excision, chemotherapy or radiation therapy, the participant has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure
* Thrombocytopenia, bleeding disorder, or anticoagulant use contraindicating intramuscular injection (a daily aspirin may be acceptable).
* Has immunosuppression as a result of an underlying illness or medications, such as antirejection/transplant regimens or immunomodulatory agents. Stable HIV disease is permitted per the following parameters:

  a. Confirmed stable HIV disease defined as documented viral load <50 copies/mL and CD4 count >200 within 6 months before enrollment, and on stable antiretroviral therapy for at least 6 months
* Has known hepatitis B (HBV) or hepatitis C (HBC). Stable HBV or HBC are permitted per the following parameters:

  1. If known HBV: confirmed inactive chronic HBV infection: HBsAg present for ≥6 months and HBeAg negative, anti-HBe positive; serum HBV DNA <2000 IU/mL; persistently normal ALT or AST levels; in those who had liver biopsy, findings that confirm absence of significant necroinflammation
  2. If known HCV: evidence of sustained virological response for ≥12 weeks after treatment or without evidence of HCV RNA viremia (undetectable HCV RNA)
* Use of oral, parenteral, or high-dose inhaled glucocorticoids*

  *For definition of high-dose inhaled glucocorticoids, reference Appendix B.
* History of Guillain-Barré syndrome
* Prior enrollment in this study during the 2021-22 flu season
* Anyone who is already enrolled or plans to enroll in another clinical trial with an investigational product during the study period.*

  *Per protocol, co-enrollment in observational or behavioral intervention studies are permitted at any time. An investigational product may be permitted for therapy of an illness condition that occurs during the study period e.g. COVID-19 illness.
* Hearing loss determined by the investigators to prevent successful communication over the phone
* History of myocarditis or pericarditis
* History of multisystem inflammatory syndrome in children (MIS-C) or adults (MIS-A).
* Has injury or other reason why deltoid site on both arms cannot be used for vaccinations.
* Any condition which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives.
* Anyone who is a relative of any research study personnel.
* Anyone who is an employee of any research study personnel.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel B Walter, MD, MPH, Principal Investigator — Duke University; Karen R Broder, MD, Principal Investigator — Centers for Disease Control and Prevention; Kawsar Talaat, MD, Principal Investigator — Johns Hopkins University; Elizabeth Schlaudecker, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - John Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walter EB, Schlaudecker EP, Talaat KR, Rountree W, Broder KR, Duffy J, Montefiori D, Poniewierski MS, Spreng RL, Staat MA, Tekalign R, Museru O, Goel A, Davis GN, Schmader KE. Immunogenicity of mRNA COVID-19 vaccine with either simultaneous or sequentially administered inactivated influenza vaccines: a randomized clinical trial. Vaccine. 2026 Feb 6;72:128072. doi: 10.1016/j.vaccine.2025.128072. Epub 2025 Dec 10. PMID 41380398
- [Derived] Walter EB, Schlaudecker EP, Talaat KR, Rountree W, Broder KR, Duffy J, Grohskopf LA, Poniewierski MS, Spreng RL, Staat MA, Tekalign R, Museru O, Goel A, Davis GN, Schmader KE. Safety of Simultaneous vs Sequential mRNA COVID-19 and Inactivated Influenza Vaccines: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2443166. doi: 10.1001/jamanetworkopen.2024.43166. PMID 39504023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 3 academic medical centers during the 2021-22 and 2022-23 flu seasons.
Pre-assignment Details: Of the 348 enrolled participants, 335 met inclusion criteria and were randomized to treatment.
Groups:
- Simultaneous Vaccination Group: Subjects will receive a dose of mRNA COVID-19 vaccine (either as a study procedure or standard of care) and IIV4 at Visit 1, saline placebo at Visit 2, and mRNA COVID-19 vaccine at Visit 3 for participants receiving their primary series of mRNA COVID-19 vaccine.
  mRNA COVID-19: ACIP-CDC recommended vaccine
  IIV4: ACIP recommended vaccine
  Placebo: Saline Control
- Sequential Vaccination Group: Subjects will receive a dose of mRNA COVID-19 vaccine (either as a study procedure or standard of care) and saline placebo at Visit 1, IIV4 at Visit 2, and mRNA COVID-19 vaccine at Visit 3 for participants receiving their primary series of mRNA COVID-19 vaccine.
  mRNA COVID-19: ACIP-CDC recommended vaccine
  IIV4: ACIP recommended vaccine
  Placebo: Saline Control
Period: Overall Study
Arm/Group | Simultaneous Vaccination Group | Sequential Vaccination Group
Started | 169 | 166
Completed | 168 | 166
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simultaneous Vaccination Group | Sequential Vaccination Group | Total
Number analyzed (Participants) | 169 | 166 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (8.0) | 33.1 (9.0) | 33.4 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 115 | 211
  Male | 73 | 51 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 156 | 156 | 312
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 15 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 30 | 60
  White | 117 | 112 | 229
  More than one race | 9 | 7 | 16
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 169 | 166 | 335

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants With Moderate or More Severe Fever, Chills, Myalgia, or Arthralgia in the Simultaneous Group and the Sequential Group Following Both Vaccination Visit 1 and 2
Description: Subjects will be asked to complete a memory aid to document symptoms and measure temperature daily.
Time Frame: Up to 7 Days Post Vaccination (combined for Visits 1 and 2)
Population: Data combined for combined for Visits 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Group | Sequential Vaccination Group
Number analyzed (Participants) | 168 | 166
Participants | 43 | 52
Statistical Analysis 1: Comparison: Simultaneous Vaccination Group vs Sequential Vaccination Group; The null hypothesis is the Simultaneous group is inferior (i.e., Simultaneous group will have a higher proportion) to the Sequential group in regards to the proportion of participants with at least one moderate or severe fever, chills, myalgia, or arthralgia event after visits 1 and 2 using 10% non-inferiority margin; Test type: Non-Inferiority — One-sided non-inferiority test with the alpha level set at 0.025 and non-inferiority margin of 10%, stratified by site; p = 0.0007, Cochran-Mantel-Haenszel — The upper limit of the 95% CI of the difference was 4% with a noninferiority margin of 10%; The upper bound of a site-stratified Newcombe binomial confidence interval with Cochran-Mantel-Haenszel weighting was used; Difference in proportions = -5.6, 95% CI 2-sided [-15.2 to 4.0]

2. Secondary Outcome: Number of Participants With Moderate or More Severe Fever, Chills, Myalgia, or Arthralgia in the Simultaneous Versus the Sequential Group Following the First Vaccination Visit
Description: Subjects will be asked to complete a memory aid to document symptoms and measure temperature daily.
Time Frame: Up to 7 Days Post Vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Group | Sequential Vaccination Group
Number analyzed (Participants) | 168 | 166
Participants | 40 | 47
Statistical Analysis 1: Comparison: Simultaneous Vaccination Group vs Sequential Vaccination Group; Test type: Superiority; p = 0.3851, Mantel Haenszel

3. Secondary Outcome: Number of Participants With Moderate or More Severe Fever, Chills, Myalgia, or Arthralgia in the Simultaneous Versus Sequential Group Following the Second Vaccination Visit
Description: Subjects will be asked to complete a memory aid to document symptoms and measure temperature daily.
Time Frame: Up to 7 Days Post Vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Group | Sequential Vaccination Group
Number analyzed (Participants) | 168 | 166
Participants | 5 | 9
Statistical Analysis 1: Comparison: Simultaneous Vaccination Group vs Sequential Vaccination Group; Test type: Superiority; p = 0.2886, Mantel Haenszel

4. Secondary Outcome: Number of Participants in the Simultaneous and Sequential Vaccination Groups With Solicited Local and Systemic Reactogenicity Events According to Severity Grade After the First, Second and Third Vaccination Visit
Description: Subjects will be asked to complete a memory aid to document symptoms and measure temperature daily.
Time Frame: Up to 7 Days Post Vaccination
Population: This study allowed participants receiving their initial two dose COVID-19 vaccine series or a COVID-19 vaccine booster to enroll. Only 4 participants were enrolled in the study who received their initial two doses of COVID-19 vaccine, and they were all randomized to the Simultaneous group. These participants received their second COVID-19 vaccine at Visit 3. Those receiving a COVID-19 booster dose did not receive any vaccine/placebo at Visit 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Group | Sequential Vaccination Group
Number analyzed (Participants) | 168 | 166
Participants
  Visit 1 Local Reaction - Pain - COVID-19 Vaccine Site: None | 39 | 27
  Visit 1 Local Reaction - Pain - COVID-19 Vaccine Site: Mild | 102 | 97
  Visit 1 Local Reaction - Pain - COVID-19 Vaccine Site: Moderate | 27 | 40
  Visit 1 Local Reaction - Pain - COVID-19 Vaccine Site: Severe | 0 | 2
  Visit 1 Local Reaction - Pain - COVID-19 Vaccine Site: Life Threatening | 0 | 0
  Visit 1 Local Reaction - Pain - Flu Vaccine/Placebo site: None | 65 | 145
  Visit 1 Local Reaction - Pain - Flu Vaccine/Placebo site: Mild | 86 | 20
  Visit 1 Local Reaction - Pain - Flu Vaccine/Placebo site: Moderate | 16 | 1
  Visit 1 Local Reaction - Pain - Flu Vaccine/Placebo site: Severe | 1 | 0
  Visit 1 Local Reaction - Pain - Flu Vaccine/Placebo site: Life Threatening | 0 | 0
  Visit 1 Local Reaction - Swelling - COVID-19 Vaccine Site: None | 164 | 156
  Visit 1 Local Reaction - Swelling - COVID-19 Vaccine Site: Mild | 4 | 4
  Visit 1 Local Reaction - Swelling - COVID-19 Vaccine Site: Moderate | 0 | 5
  Visit 1 Local Reaction - Swelling - COVID-19 Vaccine Site: Severe | 0 | 1
  Visit 1 Local Reaction - Swelling - COVID-19 Vaccine Site: Life Threatening | 0 | 0
  Visit 1 Local Reaction - Swelling - Flu Vaccine/Placebo Site: None | 164 | 164
  Visit 1 Local Reaction - Swelling - Flu Vaccine/Placebo Site: Mild | 2 | 1
  Visit 1 Local Reaction - Swelling - Flu Vaccine/Placebo Site: Moderate | 2 | 1
  Visit 1 Local Reaction - Swelling - Flu Vaccine/Placebo Site: Severe | 0 | 0
  Visit 1 Local Reaction - Swelling - Flu Vaccine/Placebo Site: Life Threatening | 0 | 0
  Visit 1 Local Reaction - Redness - COVID-19 Vaccine Site: None | 164 | 157
  Visit 1 Local Reaction - Redness - COVID-19 Vaccine Site: Mild | 4 | 6
  Visit 1 Local Reaction - Redness - COVID-19 Vaccine Site: Moderate | 0 | 2
  Visit 1 Local Reaction - Redness - COVID-19 Vaccine Site: Severe | 0 | 1
  Visit 1 Local Reaction - Redness - COVID-19 Vaccine Site: Life Threatening | 0 | 0
  Visit 1 Local Reaction - Redness - Flu Vaccine/Placebo Site: None | 165 | 165
  Visit 1 Local Reaction - Redness - Flu Vaccine/Placebo Site: Mild | 1 | 0
  Visit 1 Local Reaction - Redness - Flu Vaccine/Placebo Site: Moderate | 1 | 1
  Visit 1 Local Reaction - Redness - Flu Vaccine/Placebo Site: Severe | 1 | 0
  Visit 1 Local Reaction - Redness - Flu Vaccine/Placebo Site: Life Threatening | 0 | 0
  Visit 1 Local Reaction - Axillary - COVID-19 Vaccine Site: None | 120 | 111
  Visit 1 Local Reaction - Axillary - COVID-19 Vaccine Site: Mild | 40 | 43
  Visit 1 Local Reaction - Axillary - COVID-19 Vaccine Site: Moderate | 8 | 11
  Visit 1 Local Reaction - Axillary - COVID-19 Vaccine Site: Severe | 0 | 1
  Visit 1 Local Reaction - Axillary - COVID-19 Vaccine Site: Life Threatening | 0 | 0
  Visit 1 Local Reaction - Axillary - Flu Vaccine/Placebo Site: None | 135 | 158
  Visit 1 Local Reaction - Axillary - Flu Vaccine/Placebo Site: Mild | 29 | 5
  Visit 1 Local Reaction - Axillary - Flu Vaccine/Placebo Site: Moderate | 4 | 3
  Visit 1 Local Reaction - Axillary - Flu Vaccine/Placebo Site: Severe | 0 | 0
  Visit 1 Local Reaction - Axillary - Flu Vaccine/Placebo Site: Life Threatening | 0 | 0
  Visit 1 Systemic Reaction - Fever: None | 159 | 155
  Visit 1 Systemic Reaction - Fever: Mild | 4 | 6
  Visit 1 Systemic Reaction - Fever: Moderate | 3 | 2
  Visit 1 Systemic Reaction - Fever: Severe | 2 | 3
  Visit 1 Systemic Reaction - Fever: Life Threatening | 0 | 0
  Visit 1 Systemic Reaction - Chills: None | 121 | 116
  Visit 1 Systemic Reaction - Chills: Mild | 29 | 26
  Visit 1 Systemic Reaction - Chills: Moderate | 15 | 19
  Visit 1 Systemic Reaction - Chills: Severe | 3 | 5
  Visit 1 Systemic Reaction - Chills: Life Threatening | 0 | 0
  Visit 1 Systemic Reaction - Fatigue: None | 73 | 61
  Visit 1 Systemic Reaction - Fatigue: Mild | 50 | 61
  Visit 1 Systemic Reaction - Fatigue: Moderate | 41 | 34
  Visit 1 Systemic Reaction - Fatigue: Severe | 4 | 10
  Visit 1 Systemic Reaction - Fatigue: Life Threatening | 0 | 0
  Visit 1 Systemic Reaction - Myalgia: None | 71 | 65
  Visit 1 Systemic Reaction - Myalgia: Mild | 62 | 60
  Visit 1 Systemic Reaction - Myalgia: Moderate | 31 | 33
  Visit 1 Systemic Reaction - Myalgia: Severe | 4 | 8
  Visit 1 Systemic Reaction - Myalgia: Life Threatening | 0 | 0
  Visit 1 Systemic Reaction - Headache: None | 90 | 80
  Visit 1 Systemic Reaction - Headache: Mild | 53 | 58
  Visit 1 Systemic Reaction - Headache: Moderate | 21 | 25
  Visit 1 Systemic Reaction - Headache: Severe | 4 | 3
  Visit 1 Systemic Reaction - Headache: Life Threatening | 0 | 0
  Visit 1 Systemic Reaction - Arthralgia: None | 141 | 129
  Visit 1 Systemic Reaction - Arthralgia: Mild | 14 | 21
  Visit 1 Systemic Reaction - Arthralgia: Moderate | 12 | 11
  Visit 1 Systemic Reaction - Arthralgia: Severe | 1 | 5
  Visit 1 Systemic Reaction - Arthralgia: Life Threatening | 0 | 0
  Visit 1 Systemic Reaction - Nausea/Vomitting: None | 145 | 142
  Visit 1 Systemic Reaction - Nausea/Vomitting: Mild | 15 | 19
  Visit 1 Systemic Reaction - Nausea/Vomitting: Moderate | 7 | 3
  Visit 1 Systemic Reaction - Nausea/Vomitting: Severe | 1 | 2
  Visit 1 Systemic Reaction - Nausea/Vomitting: Life Threatening | 0 | 0
  Visit 1 Systemic Reaction - Diarrhea: None | 151 | 146
  Visit 1 Systemic Reaction - Diarrhea: Mild | 11 | 17
  Visit 1 Systemic Reaction - Diarrhea: Moderate | 6 | 2
  Visit 1 Systemic Reaction - Diarrhea: Severe | 0 | 1
  Visit 1 Systemic Reaction - Diarrhea: Life Threatening | 0 | 0
  Visit 2 Local Reaction - Pain - Flu Vaccine/Placebo Site: None | 161 | 82
  Visit 2 Local Reaction - Pain - Flu Vaccine/Placebo Site: Mild | 6 | 75
  Visit 2 Local Reaction - Pain - Flu Vaccine/Placebo Site: Moderate | 0 | 8
  Visit 2 Local Reaction - Pain - Flu Vaccine/Placebo Site: Severe | 1 | 1
  Visit 2 Local Reaction - Pain - Flu Vaccine/Placebo Site: Life Threatening | 0 | 0
  Visit 2 Local Reaction - Swelling - Flu Vaccine/Placebo Site: None | 168 | 160
  Visit 2 Local Reaction - Swelling - Flu Vaccine/Placebo Site: Mild | 0 | 4
  Visit 2 Local Reaction - Swelling - Flu Vaccine/Placebo Site: Moderate | 0 | 2
  Visit 2 Local Reaction - Swelling - Flu Vaccine/Placebo Site: Severe | 0 | 0
  Visit 2 Local Reaction - Swelling - Flu Vaccine/Placebo Site: Life Threatening | 0 | 0
  Visit 2 Local Reaction - Redness - Flu Vaccine/Placebo Site: None | 168 | 164
  Visit 2 Local Reaction - Redness - Flu Vaccine/Placebo Site: Mild | 0 | 2
  Visit 2 Local Reaction - Redness - Flu Vaccine/Placebo Site: Moderate | 0 | 0
  Visit 2 Local Reaction - Redness - Flu Vaccine/Placebo Site: Severe | 0 | 0
  Visit 2 Local Reaction - Redness - Flu Vaccine/Placebo Site: Life Threatening | 0 | 0
  Visit 2 Local Reaction - Axillary - Flu Vaccine/Placebo Site: None | 165 | 141
  Visit 2 Local Reaction - Axillary - Flu Vaccine/Placebo Site: Mild | 3 | 21
  Visit 2 Local Reaction - Axillary - Flu Vaccine/Placebo Site: Moderate | 0 | 3
  Visit 2 Local Reaction - Axillary - Flu Vaccine/Placebo Site: Severe | 0 | 1
  Visit 2 Local Reaction - Axillary - Flu Vaccine/Placebo Site: Life Threatening | 0 | 0
  Visit 2 Systemic Reaction - Fever: None | 165 | 162
  Visit 2 Systemic Reaction - Fever: Mild | 2 | 3
  Visit 2 Systemic Reaction - Fever: Moderate | 1 | 1
  Visit 2 Systemic Reaction - Fever: Severe | 0 | 0
  Visit 2 Systemic Reaction - Fever: Life Threatening | 0 | 0
  Visit 2 - Systemic Reaction - Chills: None | 167 | 157
  Visit 2 - Systemic Reaction - Chills: Mild | 0 | 7
  Visit 2 - Systemic Reaction - Chills: Moderate | 1 | 2
  Visit 2 - Systemic Reaction - Chills: Severe | 0 | 0
  Visit 2 - Systemic Reaction - Chills: Life Threatening | 0 | 0
  Visit 2 - Systemic Reaction - Fatigue: None | 150 | 121
  Visit 2 - Systemic Reaction - Fatigue: Mild | 10 | 34
  Visit 2 - Systemic Reaction - Fatigue: Moderate | 4 | 10
  Visit 2 - Systemic Reaction - Fatigue: Severe | 4 | 1
  Visit 2 - Systemic Reaction - Fatigue: Life Threatening | 0 | 0
  Visit 2 - Systemic Reaction - Myalgia: None | 159 | 124
  Visit 2 - Systemic Reaction - Myalgia: Mild | 5 | 34
  Visit 2 - Systemic Reaction - Myalgia: Moderate | 4 | 7
  Visit 2 - Systemic Reaction - Myalgia: Severe | 0 | 1
  Visit 2 - Systemic Reaction - Myalgia: Life Threatening | 0 | 0
  Visit 2 - Systemic Reaction - Headache: None | 141 | 129
  Visit 2 - Systemic Reaction - Headache: Mild | 17 | 26
  Visit 2 - Systemic Reaction - Headache: Moderate | 9 | 11
  Visit 2 - Systemic Reaction - Headache: Severe | 1 | 0
  Visit 2 - Systemic Reaction - Headache: Life Threatening | 0 | 0
  Visit 2 - Systemic Reaction - Arthralgia: None | 161 | 156
  Visit 2 - Systemic Reaction - Arthralgia: Mild | 5 | 7
  Visit 2 - Systemic Reaction - Arthralgia: Moderate | 2 | 3
  Visit 2 - Systemic Reaction - Arthralgia: Severe | 0 | 0
  Visit 2 - Systemic Reaction - Arthralgia: Life Threatening | 0 | 0
  Visit 2 - Systemic Reaction - Nausea/Vomiting: None | 163 | 160
  Visit 2 - Systemic Reaction - Nausea/Vomiting: Mild | 4 | 4
  Visit 2 - Systemic Reaction - Nausea/Vomiting: Moderate | 1 | 2
  Visit 2 - Systemic Reaction - Nausea/Vomiting: Severe | 0 | 0
  Visit 2 - Systemic Reaction - Nausea/Vomiting: Life Threatening | 0 | 0
  Visit 2 - Systemic Reaction - Diarrhea: None | 163 | 152
  Visit 2 - Systemic Reaction - Diarrhea: Mild | 5 | 14
  Visit 2 - Systemic Reaction - Diarrhea: Moderate | 0 | 0
  Visit 2 - Systemic Reaction - Diarrhea: Severe | 0 | 0
  Visit 2 - Systemic Reaction - Diarrhea: Life Threatening | 0 | 0
  Visit 3 - Local Reaction - Pain - COVID-19 Vaccine: number analyzed (Participants) | 4 | 0
  Visit 3 - Local Reaction - Pain - COVID-19 Vaccine: None | 4 | 0
  Visit 3 - Local Reaction - Pain - COVID-19 Vaccine: Mild | 0 | 0
  Visit 3 - Local Reaction - Pain - COVID-19 Vaccine: Moderate | 0 | 0
  Visit 3 - Local Reaction - Pain - COVID-19 Vaccine: Severe | 0 | 0
  Visit 3 - Local Reaction - Pain - COVID-19 Vaccine: Life Threatening | 0 | 0
  Visit 3 - Local Reaction - Swelling - COVID-19 Vaccine: number analyzed (Participants) | 4 | 0
  Visit 3 - Local Reaction - Swelling - COVID-19 Vaccine: None | 4 | 0
  Visit 3 - Local Reaction - Swelling - COVID-19 Vaccine: Mild | 0 | 0
  Visit 3 - Local Reaction - Swelling - COVID-19 Vaccine: Moderate | 0 | 0
  Visit 3 - Local Reaction - Swelling - COVID-19 Vaccine: Severe | 0 | 0
  Visit 3 - Local Reaction - Swelling - COVID-19 Vaccine: Life Threatening | 0 | 0
  Visit 3 - Local Reaction - Redness - COVID-19 Vaccine: number analyzed (Participants) | 4 | 0
  Visit 3 - Local Reaction - Redness - COVID-19 Vaccine: None | 4 | 0
  Visit 3 - Local Reaction - Redness - COVID-19 Vaccine: Mild | 0 | 0
  Visit 3 - Local Reaction - Redness - COVID-19 Vaccine: Moderate | 0 | 0
  Visit 3 - Local Reaction - Redness - COVID-19 Vaccine: Severe | 0 | 0
  Visit 3 - Local Reaction - Redness - COVID-19 Vaccine: Life Threatening | 0 | 0
  Visit 3 - Local Reaction - Axillary - COVID-19 Vaccine: number analyzed (Participants) | 4 | 0
  Visit 3 - Local Reaction - Axillary - COVID-19 Vaccine: None | 3 | 0
  Visit 3 - Local Reaction - Axillary - COVID-19 Vaccine: Mild | 1 | 0
  Visit 3 - Local Reaction - Axillary - COVID-19 Vaccine: Moderate | 0 | 0
  Visit 3 - Local Reaction - Axillary - COVID-19 Vaccine: Severe | 0 | 0
  Visit 3 - Local Reaction - Axillary - COVID-19 Vaccine: Life Threatening | 0 | 0
  Visit 3 - Systemic Reaction - Fever: number analyzed (Participants) | 4 | 0
  Visit 3 - Systemic Reaction - Fever: None | 4 | 0
  Visit 3 - Systemic Reaction - Fever: Mild | 0 | 0
  Visit 3 - Systemic Reaction - Fever: Moderate | 0 | 0
  Visit 3 - Systemic Reaction - Fever: Severe | 0 | 0
  Visit 3 - Systemic Reaction - Fever: Life Threatening | 0 | 0
  Visit 3 - Systemic Reaction - Chills: number analyzed (Participants) | 4 | 0
  Visit 3 - Systemic Reaction - Chills: None | 4 | 0
  Visit 3 - Systemic Reaction - Chills: Mild | 0 | 0
  Visit 3 - Systemic Reaction - Chills: Moderate | 0 | 0
  Visit 3 - Systemic Reaction - Chills: Severe | 0 | 0
  Visit 3 - Systemic Reaction - Chills: Life Threatening | 0 | 0
  Visit 3 - Systemic Reaction - Fatigue: number analyzed (Participants) | 4 | 0
  Visit 3 - Systemic Reaction - Fatigue: None | 3 | 0
  Visit 3 - Systemic Reaction - Fatigue: Mild | 1 | 0
  Visit 3 - Systemic Reaction - Fatigue: Moderate | 0 | 0
  Visit 3 - Systemic Reaction - Fatigue: Severe | 0 | 0
  Visit 3 - Systemic Reaction - Fatigue: Life Threatening | 0 | 0
  Visit 3 - Systemic Reaction - Myalgia: number analyzed (Participants) | 4 | 0
  Visit 3 - Systemic Reaction - Myalgia: None | 4 | 0
  Visit 3 - Systemic Reaction - Myalgia: Mild | 0 | 0
  Visit 3 - Systemic Reaction - Myalgia: Moderate | 0 | 0
  Visit 3 - Systemic Reaction - Myalgia: Severe | 0 | 0
  Visit 3 - Systemic Reaction - Myalgia: Life Threatening | 0 | 0
  Visit 3 - Systemic Reaction - Headache: number analyzed (Participants) | 4 | 0
  Visit 3 - Systemic Reaction - Headache: None | 3 | 0
  Visit 3 - Systemic Reaction - Headache: Mild | 1 | 0
  Visit 3 - Systemic Reaction - Headache: Moderate | 0 | 0
  Visit 3 - Systemic Reaction - Headache: Severe | 0 | 0
  Visit 3 - Systemic Reaction - Headache: Life Threatening | 0 | 0
  Visit 3 - Systemic Reaction - Arthralgia: number analyzed (Participants) | 4 | 0
  Visit 3 - Systemic Reaction - Arthralgia: None | 4 | 0
  Visit 3 - Systemic Reaction - Arthralgia: Mild | 0 | 0
  Visit 3 - Systemic Reaction - Arthralgia: Moderate | 0 | 0
  Visit 3 - Systemic Reaction - Arthralgia: Severe | 0 | 0
  Visit 3 - Systemic Reaction - Arthralgia: Life Threatening | 0 | 0
  Visit 3 - Systemic Reaction - Nausea/Vomiting: number analyzed (Participants) | 4 | 0
  Visit 3 - Systemic Reaction - Nausea/Vomiting: None | 3 | 0
  Visit 3 - Systemic Reaction - Nausea/Vomiting: Mild | 1 | 0
  Visit 3 - Systemic Reaction - Nausea/Vomiting: Moderate | 0 | 0
  Visit 3 - Systemic Reaction - Nausea/Vomiting: Severe | 0 | 0
  Visit 3 - Systemic Reaction - Nausea/Vomiting: Life Threatening | 0 | 0
  Visit 3 - Systemic Reaction - Diarrhea: number analyzed (Participants) | 4 | 0
  Visit 3 - Systemic Reaction - Diarrhea: None | 4 | 0
  Visit 3 - Systemic Reaction - Diarrhea: Mild | 0 | 0
  Visit 3 - Systemic Reaction - Diarrhea: Moderate | 0 | 0
  Visit 3 - Systemic Reaction - Diarrhea: Severe | 0 | 0
  Visit 3 - Systemic Reaction - Diarrhea: Life Threatening | 0 | 0

5. Secondary Outcome: Number of Participants With Observed Serious Adverse Events
Time Frame: 120 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Group | Sequential Vaccination Group
Number analyzed (Participants) | 169 | 166
Participants | 1 | 1
Statistical Analysis 1: Comparison: Simultaneous Vaccination Group vs Sequential Vaccination Group; Test type: Other; The comparison in number of participants with reported SAEs regardless of relationship to study product were made using a difference in proportions along with a 95% confidence interval of the difference; Comparison of Frequencies = -0.01, 95% CI 2-sided [-1.66 to 1.64]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 120 days (approximately 4 months).
Arm/Group | Simultaneous Vaccination Group | Sequential Vaccination Group
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/166
Serious Adverse Events (participants affected / at risk) | 1/169 | 1/166
Other Adverse Events (participants affected / at risk) | 18/169 | 9/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous Vaccination Group (N=169) | Sequential Vaccination Group (N=166)
Spontaneous Complete Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous Vaccination Group (N=169) | Sequential Vaccination Group (N=166)
COVID-19 Illness (Infections and infestations) | 18 (18) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT05028361/Prot_003.pdf
  • Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT05028361/SAP_004.pdf
  • Informed Consent Form (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT05028361/ICF_002.pdf